CLINICAL TRIAL: NCT07123064
Title: Alleviating Loneliness in Older Adults Living in Poverty: A Multi-level Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: University College, London (Other); The Hong Kong Polytechnic University (Other); University of Texas at Austin (Other); Australian National University (Other); The University of Hong Kong (Other); Medical School Berlin (Other); Chinese University of Hong Kong (Other); University of Bern (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Chou Kee Lee, Chair Professor of Social Policy, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-2024-0624; R8002-24 (Other Grant/Funding Number: Research Impact Fund, Research Grants Council)
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Loneliness; Poverty
Keywords: Loneliness; Poverty; Cluster Randomized Controlled Trials; Older Adults; Mindfulness; SOLUS-D Programme; Group 4 Health; Neighbour Every Day; Hong Kong

STUDY DESIGN:
Intervention Model Description: Single Blinded, 4-arm cluster randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First Arm (Experimental): Individual-level
  Interventions: Behavioral: Individual Level
- Second Arm (Experimental): Individual- and Interpersonal-level
  Interventions: Behavioral: Individual Level; Behavioral: Interpersonal Level
- Third Arm (Experimental): Individual-, Interpersonal-, and Community-level
  Interventions: Behavioral: Individual Level; Behavioral: Interpersonal Level; Behavioral: Community Level
- Forth Arm (Active Comparator): Education Control Group
  Interventions: Other: Education Control

INTERVENTIONS:
Behavioral: Individual Level — A 8-weekly, 1hour telephone-delivered sessions using mindfulness and SOLUS-D program. Key contents include: introduction to mindfulness - Body awareness and present moment experiences, emotional awareness and mind-body labeling, relaxation techniques and sensory discrimination, deepening awareness and accepting feelings, personal values, interconnection between thought patterns and emotions, identifying and analyzing of thought traps, and challenging thoughts and future planning. Maintenance sessions which focus on embedding mindfulness practices and SOLUS-D program among older adults as a persistent habit will be conducted.
  Arms: First Arm; Second Arm; Third Arm
Behavioral: Interpersonal Level — A 8 weekly, 1hr sessions through telephone or Zoom using the Group 4 Health. Key contents include: understanding the benefits of social connections, exploring self and community, community and action, support and breakthrough, summary and moving forward. Maintenance sessions which focus on continuous practice of support and community will be conducted.
  Arms: Second Arm; Third Arm
Behavioral: Community Level — A 4 weekly, 2hour in-person sessions through (1) strengthening collective efficacy via neighbor identification with the community. Key contents include: building neighbourhood connections, getting to know each other, health aging, neighbourhood care, vibrant exploration, thriving community, connecting the dots.
  Arms: Third Arm
Other: Education Control — Monthly monthly messages via text, graphics or voice recordings will be sent over a period of 6 months. Key content includes: healthy diet tips, recognizing warning signs of health, understanding dementia, fall prevention tips, health message, and anti-fraud tips.
  Arms: Forth Arm

SUMMARY:
The study aims to reduce loneliness among Hong Kong Chinese older adults living in poverty with a multi-level intervention involving components at the individual, interpersonal, and community levels.

DETAILED DESCRIPTION:
Loneliness is widespread, with negative impacts on both individuals and society and associated direct and indirect healthcare and long-term care costs. Thus, it is imperative to alleviate loneliness in old age by implementing effective, accessible, affordable, and scalable interventions. Loneliness is often erroneously considered an individual problem due to personal failure. Still, growing evidence indicates that loneliness is caused by factors at multiple levels, including the individual, interpersonal, and community levels. Hence, a multi-level approach is recommended to alleviate loneliness.

However, multi-level interventions for reducing loneliness are in their infancy, and there is yet to be evidence to suggest that they are more effective than single-level interventions. The investigators will conduct an innovative and impactful study to fill this important research gap. This study is a single-blinded cluster, four-arm randomized controlled trial (RCT) designed to test the effect and cost-effectiveness of a multi-level intervention to alleviate loneliness among Hong Kong Chinese older adults living in poverty. The investigators will also adopt the modified biopsychosocial (BPS) model, called the BPS-Pathways model, as the theoretical framework to guide our selection of interventions, mediators, secondary outcomes, long-term outcomes, and impact.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older
* living in poverty (defined: inability to afford at least 5 items on the material deprivation index)
* proficiency in spoken Cantonese
* experiencing loneliness (defined: score of ≥ 6 on the 3-item UCLA Loneliness Scale)

Exclusion Criteria:

* cognitive impairments, psychiatric disorders, learning disabilities, or active suicidal ideation
* actively participating in other psychotherapy or psychosocial interventions in the past 1 year

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1344 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
UCLA Loneliness Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  The 20-item UCLA Loneliness Scale is a reliable self-assessment tool designed to evaluate feelings of loneliness. Each item will be rated from 1=Never to 4=Always. Total scores range from 20 to 80.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  PSQI evaluates seven components of sleep: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction. Each item will be rated from 0=No difficulty to 3=Severe difficulty. Total scores range from 0 to 21,
Satisfaction with Life Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  SWLS measures the subjective well-being and life satisfaction. Each item will be rated from 1=Strongly disagree to 7=Strongly agree. Total scores range from 5 to 35.
De Jong Gierveld Loneliness Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  The De Jong Gierveld Loneliness Scale is known for assessing loneliness with social and emotional loneliness subscale. Each item will be rated from 1=Yes to 3=No. Total scores range from 0 to 6, with subscale score ranging from 0 to 3.
Lawton Instrumental Activities of Daily Living | Baseline, 12-month, 24-month
  IADL is used to measure participant's ability in performing instrumental activities. Each item will be rated 0=dependent to 1=independent. Total scores range from 0 to 8.
Activities of Daily Living | Baseline, 12-month, 24-month
  ADL is used to measure participant's independence in completing activities of daily living. Each item will be rate from 0=dependent to 5/10=independent. Total scores range from 0 to 100.
Physical Symptoms Inventory | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  Participants will rate the presence of each physical symptom in the past 30 days from 0=Never to 4=Often. Total scores range from 0 to 72.
Charlson Comorbidity Index | Baseline, 12-month, 24-month
  Participants will rate the presence a list of 16 comorbid condition. Total scores range from 0 to 37.
Perceived Stress Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  PSS is use to measure perceived stress levels. Each item will be rated from 0=Never to 4=Very often. Total scores range from 0 to 56.
6-Minutes Walking Test | Baseline, 12-month, 24-month
  Participants will be asked to walk the furthest distance possible in 6 minutes, rate their level of breathlessness using the Borg scale from 0=No breathlessness to 10=Maximal breathlessness.
Hospital Anxiety and Depression Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  HADS measure the severity of anxiety and depression. Each item will be rated from 0=Not at all to 3=Most of the time. Total score range from 0 to 42.
Montreal Cognitive Assessment - Hong Kong | Baseline, 12-month, 24-month
  MoCA-HK is a tool to evaluate cognitive functioning in older adults, which compromises of seven cognitive domains. Total score range from 0 to 30.

OTHER OUTCOMES:
Mindfulness Attention Awareness Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  Each item will be rated from 1=Almost always to 6=Almost never. Average score will be calculated.
Self-Compassion Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  SCS-SF measures self-compassion and have 6 subscales. Each item will be rated from 1=Almost never to 5=Almost always. Mean score will be calculated for each subscale and overall scale.
Emotion Regulation Questionnaire | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  ERQ-CR is used for assessing emotional regulation strategies; cognitive reappraisal (6 items). Each item will be rated from 1=Strongly disagree to 7=Strongly agree. Mean score will be calculated.
Multidimensional Scale of Perceived Social Support | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  MSPSS evaluates the social support derived from three key sources: family, friends, and significant others. Each item will be rated from 1=Strongly disagree to 7=Strongly agree. Total scores range from 12 to 84.
Lubben Social Network Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  LSNS is used to assess the social networks of participants. Each item will be rated 0=None to 5=9 or more. Total scores range from 0 to 30.
Neighbourhood Collective Efficacy Scale | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  NEC assesses the neighborhood collective efficacy and identity of the community. Each item will be rated from from 1=Strongly agree to 5=Strongly disagree. Mean score will be calculated.
EuroQol 5-dimension 5-level instrument | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  EQ-5D-5L assesses descriptive system and visual analogue scale. Participants will rate their health status from 0=No problem to 5=Unable to perform, and their overall health status on the day of assessment from 0=Worst health to 100=Best health.
Healthcare Service Usage | Baseline, 2-month, 4-month, 6-month, 12-month, 24-month
  Participants will rate their frequency of use of outpatient medical treatment, accident and emergency treatment, and inpatient medical treatment over the past three months at both public and private facilities from 0=None to 3=three times or more.

CONTACTS AND LOCATIONS:
Overall Officials: Kee Lee Chou, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Surkalim DL, Luo M, Eres R, Gebel K, van Buskirk J, Bauman A, Ding D. The prevalence of loneliness across 113 countries: systematic review and meta-analysis. BMJ. 2022 Feb 9;376:e067068. doi: 10.1136/bmj-2021-067068. PMID 35140066
- [Background] Seguin-Fowler RA, Graham ML, Demment M, Uribe ALM, Rethorst CD, Szeszulski J. Multilevel Interventions Targeting Obesity: State of the Science and Future Directions. Annu Rev Nutr. 2024 Aug;44(1):357-381. doi: 10.1146/annurev-nutr-122123-020340. Epub 2024 Aug 12. PMID 38885446
- [Background] Santini ZI, Koyanagi A, Tyrovolas S, Haro JM, Fiori KL, Uwakwa R, Thiyagarajan JA, Webber M, Prince M, Prina AM. Social network typologies and mortality risk among older people in China, India, and Latin America: A 10/66 Dementia Research Group population-based cohort study. Soc Sci Med. 2015 Dec;147:134-43. doi: 10.1016/j.socscimed.2015.10.061. Epub 2015 Nov 4. PMID 26575604
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Masi CM, Chen HY, Hawkley LC, Cacioppo JT. A meta-analysis of interventions to reduce loneliness. Pers Soc Psychol Rev. 2011 Aug;15(3):219-66. doi: 10.1177/1088868310377394. Epub 2010 Aug 17. PMID 20716644
- [Background] Lloyd-Evans B, Frerichs J, Stefanidou T, Bone J, Pinfold V, Lewis G, Billings J, Barber N, Chhapia A, Chipp B, Henderson R, Shah P, Shorten A, Giorgalli M, Terhune J, Jones R, Johnson S. The Community Navigator Study: Results from a feasibility randomised controlled trial of a programme to reduce loneliness for people with complex anxiety or depression. PLoS One. 2020 May 29;15(5):e0233535. doi: 10.1371/journal.pone.0233535. eCollection 2020. PMID 32469922
- [Background] Lengnick-Hall R, Williams NJ, Ehrhart MG, Willging CE, Bunger AC, Beidas RS, Aarons GA. Eight characteristics of rigorous multilevel implementation research: a step-by-step guide. Implement Sci. 2023 Oct 23;18(1):52. doi: 10.1186/s13012-023-01302-2. PMID 37872618
- [Background] Hunter RF, de la Haye K, Murray JM, Badham J, Valente TW, Clarke M, Kee F. Social network interventions for health behaviours and outcomes: A systematic review and meta-analysis. PLoS Med. 2019 Sep 3;16(9):e1002890. doi: 10.1371/journal.pmed.1002890. eCollection 2019 Sep. PMID 31479454
- [Background] Hickin N, Kall A, Shafran R, Sutcliffe S, Manzotti G, Langan D. The effectiveness of psychological interventions for loneliness: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Aug;88:102066. doi: 10.1016/j.cpr.2021.102066. Epub 2021 Jul 18. PMID 34339939
- [Background] Harada K, Masumoto K, Katagiri K, Fukuzawa A, Touyama M, Sonoda D, Chogahara M, Kondo N, Okada S. Three-year effects of neighborhood social network intervention on mental and physical health of older adults. Aging Ment Health. 2021 Dec;25(12):2235-2245. doi: 10.1080/13607863.2020.1839858. Epub 2020 Oct 29. PMID 33118392
- [Background] Fong P, Cruwys T, Robinson SL, Haslam SA, Haslam C, Mance PL, Fisher CL. Evidence that loneliness can be reduced by a whole-of-community intervention to increase neighbourhood identification. Soc Sci Med. 2021 May;277:113909. doi: 10.1016/j.socscimed.2021.113909. Epub 2021 Apr 6. PMID 33866082
- [Background] Ernst M, Niederer D, Werner AM, Czaja SJ, Mikton C, Ong AD, Rosen T, Brahler E, Beutel ME. Loneliness before and during the COVID-19 pandemic: A systematic review with meta-analysis. Am Psychol. 2022 Jul-Aug;77(5):660-677. doi: 10.1037/amp0001005. Epub 2022 May 9. PMID 35533109
- [Background] Cruwys T, Fong P, Evans O, Rathbone JA. A community-led intervention to build neighbourhood identification predicts better wellbeing following prolonged COVID-19 lockdowns. Front Psychol. 2022 Dec 9;13:1030637. doi: 10.3389/fpsyg.2022.1030637. eCollection 2022. PMID 36571042
- [Background] Creswell JD, Irwin MR, Burklund LJ, Lieberman MD, Arevalo JM, Ma J, Breen EC, Cole SW. Mindfulness-Based Stress Reduction training reduces loneliness and pro-inflammatory gene expression in older adults: a small randomized controlled trial. Brain Behav Immun. 2012 Oct;26(7):1095-101. doi: 10.1016/j.bbi.2012.07.006. Epub 2012 Jul 20. PMID 22820409
- [Background] Chung GK, Robinson M, Marmot M, Woo J. Monitoring socioeconomic inequalities in health in Hong Kong: insights and lessons from the UK and Australia. Lancet Reg Health West Pac. 2022 Nov 11;31:100636. doi: 10.1016/j.lanwpc.2022.100636. eCollection 2023 Feb. PMID 36879790
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Agurs-Collins T, Persky S, Paskett ED, Barkin SL, Meissner HI, Nansel TR, Arteaga SS, Zhang X, Das R, Farhat T. Designing and Assessing Multilevel Interventions to Improve Minority Health and Reduce Health Disparities. Am J Public Health. 2019 Jan;109(S1):S86-S93. doi: 10.2105/AJPH.2018.304730. PMID 30699029